CLINICAL TRIAL: NCT06526598
Title: A Cluster Randomized Trial on Inspiratory Effort-Based Pressure Support Adjustment Strategy in Patients Undergoing Assisted Mechanical Ventilation
Brief Title: Inspiratory Effort-Targeted Pressure Support Ventilation (IT-PSV) Trial
Acronym: IT-PSV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT2024-029-004
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Critical Care; Acute Hypoxic Respiratory Failure; Ventilator-Induced Lung Injury
Keywords: pressure support ventilation; pressure muscle index; inspiratory effort
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMI-targeted group (Experimental): The participants will be treated according to the standard of care for mechanical ventilation. During PSV, pressure support is set and adjusted according to the PMI target.
  Interventions: Procedure: PMI-targeted pressure support setting and adjustment
- VT/RR-targeted group (Active Comparator): The participants will be treated according to the standard of care for mechanical ventilation. During PSV, pressure support is set and adjusted according to the VT/RR target.
  Interventions: Procedure: VT/RR-targeted pressure support setting and adjustment

INTERVENTIONS:
Procedure: PMI-targeted pressure support setting and adjustment — During PSV, the pressure support is set and adjusted to a PMI target between 0 and 2 cmH2O.
  Arms: PMI-targeted group
Procedure: VT/RR-targeted pressure support setting and adjustment — During PSV, pressure support is set and adjusted according to a VT/RR target of VT between 6 and 8 ml/kg predicted body weight, RR between 20 and 35 breaths/min, and no signs of respiratory distress.
  Arms: VT/RR-targeted group

SUMMARY:
The Inspiratory effort-Targeted Pressure Support Ventilation (IT-PSV) is a cluster randomized controlled trial. Its main aim is to determine whether an inspiratory effort-targeted pressure support setting strategy, compared to the traditional tidal volume and respiratory rate target, can improve clinical outcomes in adult participants undergoing pressure support ventilation.

The investigators propose a physiological-oriented assisted ventilation management that, if found effective, could potentially change the clinical practice for mechanical ventilation.

DETAILED DESCRIPTION:
Pressure-support ventilation (PSV) is widely used in the intensive care unit (ICU). The successful implementation of PSV depends on matching the patient's inspiratory effort with the ventilator support. Traditionally, pressure support levels are set according to tidal volume (VT) and respiratory rate (RR). However, previous studies have shown that over-assistance under PSV is not uncommon based on this setting strategy. Pressure muscle index (PMI) is an inspiratory effort monitoring, which can be easily obtained on the ventilator screen at the bedside.

Aim:

The aim is to determine whether an inspiratory effort-targeted pressure support setting strategy, compared to the traditional approach, can improve clinical outcomes in adult participants undergoing PSV.

Design:

This is a two-arm cluster randomized trial in 18 clusters randomized 1:1 to pressure support setting by a PMI-targeted strategy or a traditional VT/RR-targeted strategy.

Population:

Patients with acute hypoxic respiratory failure who have been intubated within seven days and undergoing PSV within 24 hours will be enrolled.

Intervention:

During the study, a general standard of care for mechanical ventilation will be followed, including the transition of control modes to PSV, the principle PSV settings (trigger, cycle-off, fraction of inspired oxygen, and positive end-expiratory pressure), rescue backup of controlled ventilation, performance of spontaneous breathing trial, and weaning and extubation.

In the VT/RR-targeted group, the pressure support is adjusted to obtain a VT between 6 and 8 ml/kg predicted body weight and RR between 20 and 35 breaths/min.

In the PMI-targeted group, the pressure support is adjusted according to the PMI between 0 and 2 cmH2O.

During the study period in the two groups, pressure support adjustment will be performed at least twice daily.

The intervention will be implemented over 24 months.

Training:

After randomization, a four-week comprehensive training program will be conducted for all staff in the participating ICUs before the formal start of the trial.

Outcomes:

The primary outcome is the ventilator free day during 28 days. Secondary outcomes include total duration of mechanical ventilation, the time before the first spontaneous breathing trial, weaning time, frequency of prolonged and failed weaning, frequency of mechanical ventilation longer than 21 days, length of stay in the ICU and hospital, ICU mortality, hospital mortality, and 28-day mortality.

Study sites:

The study will be conducted in 18 ICUs in university-affiliated hospitals in three provinces in China: Beijing, Tianjin, and Hebei.

ELIGIBILITY:
Mechanically ventilated patients, who are admitted to the ICU with acute hypoxic respiratory failure, will be consecutively screened daily at 08:00-10:00 morning rounds.

Inclusion criteria:

1. PSV initiated during the last 24 hours;
2. Mechanical ventilation expected to be required for at least 24-48 h by responsible physicians;
3. The partial pressure of oxygen in arterial blood (PaO2)/inspired oxygen fraction (FiO2) ≤ 300 mmHg (measuring at clinical FiO2 and positive end-expiratory pressure PEEP);
4. No sedation or stable sedation with Richmond Agitation Sedation Scale (RASS) of -2 to +1 or Riker's Sedation-Agitation Scale (SAS) of 3 to 4.

Exclusion criteria included:

1. Age younger than 18 years old;
2. Initiation of PSV before ICU admission;
3. Duration of mechanical ventilation longer than 7 days before enrollment;
4. History of neuromuscular diseases;
5. Clinical suspicion of increased intracranial pressure;
6. Extracorporeal support;
7. Moribund conditions;
8. Refusal by the ICU physicians or the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days (VFDs) at day 28 after enrollment. | 28 days
  The primary outcome is the ventilator-free days (VFDs) at day 28 after enrollment. The calculation of VFDs will follow the standard recommendations.

SECONDARY OUTCOMES:
Duration of mechanical ventilation after enrollment | 28 days
  Defined as the time intervals from enrollment to successful weaning. For patients with re-intubation or restoration of mechanical ventilation via tracheostomy within seven days after extubation and discontinuation of ventilation, the thereafter duration will be added.
The time before the first spontaneous breathing trial | 28 days
  Defined as the time interval from intubation and mechanical ventilation to the first spontaneous breathing trial attempt.
Weaning time | 28 days
  Defined as the time from the first SBT attempt to successful discontinuation of mechanical ventilation.
Frequency of prolonged weaning | 28 days
  Prolonged weaning is defined as that weaning is still not terminated 7 days after the first separation attempt.
ICU mortality | 28 days
  Death in the ICU.
Hospital mortality | 28 days
  Death in the hospital.
Length of stay in the ICU | 28 days
  Defined as the time interval from enrollment to discharge from ICU or death.
Length of stay in the hospital | 28 days
  Defined as the time interval from enrollment to discharge from hospital or death.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Shijitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu WY, Miao MY, Gao R, Yang YL, Zhang L, Weng L, Zhu FX, Liu L, Zhou JX. A cluster randomized trial on inspiratory effort-targeted pressure support adjustment strategy in patients undergoing assisted mechanical ventilation: protocol for the IT-PSV study. Front Med (Lausanne). 2024 Nov 8;11:1483976. doi: 10.3389/fmed.2024.1483976. eCollection 2024. PMID 39582975